CLINICAL TRIAL: NCT00306865
Title: Evaluation of Density and Pattern of Distribution of GABA A Receptors in the Brain of Patients With Focal Hand Dystonia Studied With PET Using [11C] Flumazenil
Brief Title: Brain Changes in Patients With Focal Hand Dystonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060031; 06-N-0031
Record Dates: First submitted 2006-03-23; First posted 2006-03-24 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-10-14

CONDITIONS: Focal Dystonia
Keywords: Neurotransmitter; Neuroimaging; Movement Disorder; Focal Hand Dystonia; FHD; HV
MeSH Terms: conditions — Dystonic Disorders; Movement Disorders; Dystonia, Focal, Task-Specific

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will examine how chemical changes in the brain produce symptoms of hand dystonia. Patients with dystonia have muscle spasms that cause uncontrolled twisting and repetitive movement or abnormal postures. In focal dystonia, just one part of the body, such as the hand, neck or face, is involved. The study will use positron emission tomography (PET) to find our which areas of the brain in patients with focal hand dystonia differ from healthy volunteers without focal hand dystonia.

Healthy volunteers and patients with focal hand dystonia between 18 and 65 years of age may be eligible for this study. Candidates are screened with a medical history and physical and neurological examinations.

Participants undergo the following procedures:

* PET scanning: The PET scanner is shaped like a doughnut. The subject lies on a bed that can slide in and out of the scanner. A custom-molded plastic mask is placed on the face and head to support the head and prevent it from moving during scanning. Two radioactive substances - five doses (one per scan) of [15 O] water and one dose of [11C] flumazil are injected into the body through a vein. The dose of injected radioactive substance is very small, and they are not harmful to the body. The [15 O] water doses are injected during the first hour and scans are taken every 10 minutes. The [11C] flumazil is injected during the second hour. The radioactive substances are detected by the PET scanner and provide information on the functioning of the brain chemistry.
* MRI scanning: MRI uses a magnetic field and radio waves to produce images of body tissues and organs. The patient lies on a table that is moved into the scanner (a narrow cylinder), wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. Scanning time for this study will be less than one hour. Subjects may be asked to lie still for up to 10 minutes at a time.

DETAILED DESCRIPTION:
Objective

The purpose of this study is to determine if in focal hand dystonia there is disinhibition involving key structures of the motor control system (basal ganglia, thalamus, cerebellum and motor cortex) caused by dysfunction of the GABA-ergic neurons. The major inhibitory neurotransmitter in the central nervous system is gamma-amino butyric acid (GABA), which acts mainly through GABA A receptors, the majority of which possess the benzodiazepine binding site. Pathological processes involving GABA-ergic neurons will cause alterations in the density of GABA receptors, which can be visualized and measured with positron emission tomography (PET) using as a radioactive ligand [(11)C] Flumazenil.

Study Population

This research will be conducted using 20 patients with primary focal hand dystonia and 20 healthy volunteers that are matched by age and gender.

Design

By using positron emission tomography (PET) using radioactive ligand [(11)C] Flumazenil, we will detect alterations in the density of GABA receptors in patients with primary focal hand dystonia in comparison with control subjects.

Outcome Measures

We will be able to determine the density of GABA A receptors of the various Regions of Interest as measured by PET analysis among these groups of subjects. This study should provide new information concerning localization and degree of dysfunction of GABA-ergic neurons in movement related structures in dystonia, which might open new possibilities for pharmacological treatment of this disorder.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Patients will have clinically documented focal hand dystonia. This criterion will be established by the preliminary screening in the NINDS Human Motor Control Section Outpatient Clinic.

B. Patients (male or female) will range in age from 18 through 65 years of age. Female patients of childbearing potential will have a pregnancy test, which must be negative and an interview prior to the study to ensure that pregnant patients do not participate in the study. Subjects will be asked to abstain from alcohol for one week prior to the study.

C. Twenty healthy volunteers will be included; volunteers will be screened in the NINDS Human Motor Control Section Outpatient Clinic, and will have neurological and physical examinations. Healthy volunteers with chronic illnesses, taking any medication that affects the CNS will be excluded. Subjects will be asked to abstain from alcohol for one week prior to the study. Female volunteers of childbearing potential will have a pregnancy test, which must be negative and an interview prior to the study to ensure that pregnant subjects do not participate in the study.

EXCLUSION CRITERIA:

The following subjects will be excluded:

A. Subjects younger than 18 and older than 65 years old.

B. Subjects with MRI findings consistent with brain tumors, strokes, trauma or AVMs.

C. Patients with progressive neurological disorders other than dystonia.

D. Subjects with past or present neuropsychiatric illness, head trauma with loss of consciousness, epilepsy, cerebro-vascular disease, migraine, past and present history of alcohol abuse, medical conditions that may alter cerebral structure.

E. Subjects with cancer, except for skin cancer.

F. Subjects incapable of giving an informed consent

G. Subjects who are pregnant or breastfeeding

H. Patients who are currently on benzodiazepines, which binds GABA-A receptors and will compete directly with flumazenil for binding; baclofen which binds GABA-B receptors; flunitrazepam, a benzodiazepine receptor agonist; or triazolam, a partial allosteric modulator of GABA A receptors. Patients need to be off of these medications for four weeks prior to entering the study.

I. Patients who have had recent (within 3 months) BoTox injections. Botulinum Toxin A (BoTox) injections are commonly used to relieve pain and muscle spasms of dystonic patients.

Participation of Children

Patients or healthy subjects younger than 18 years of age will be excluded from the study due to the following reasons:

(i) Absorbed radiation dose per mCi is relatively higher, and pharmacodynamic effects are greater in children compared to adults. (ii) No direct benefit for individual patients is anticipated from this study. The study is of "greater than minimal risk", and thus does not meet the criterion of 45 CFR 46 Subpart D (the "prospect of direct benefit") governing participation of children in research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-03-17; Study Completion 2010-10-14

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bara-Jimenez W, Catalan MJ, Hallett M, Gerloff C. Abnormal somatosensory homunculus in dystonia of the hand. Ann Neurol. 1998 Nov;44(5):828-31. doi: 10.1002/ana.410440520. PMID 9818942
- [Background] Bennett BD, Bolam JP. Localisation of parvalbumin-immunoreactive structures in primate caudate-putamen. J Comp Neurol. 1994 Sep 15;347(3):340-56. doi: 10.1002/cne.903470303. PMID 7822489
- [Background] Bolam JP, Hanley JJ, Booth PA, Bevan MD. Synaptic organisation of the basal ganglia. J Anat. 2000 May;196 ( Pt 4)(Pt 4):527-42. doi: 10.1046/j.1469-7580.2000.19640527.x. PMID 10923985